CLINICAL TRIAL: NCT05855486
Title: An Interventional, Non-comparative, Single-center Post Marketing Clinical Follow-up (PMCF) Study to Evaluate Performance and Safety of "LUXIDROPIN BABY & JUNIOR" Used to Facilitate the Removal of Ocular Secretions in Pediatric Subjects
Brief Title: PMCF Study to Evaluate Performance and Safety of "LUXIDROPIN BABY & JUNIOR"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C.O.C. Farmaceutici S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COC-R7-BABY
Record Dates: First submitted 2023-04-13; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Ocular Discharge

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eyedrops treatment arm (Experimental)
  Interventions: Device: Saline eye drops

INTERVENTIONS:
Device: Saline eye drops — Ocular drops used to facilitate the removal of ocular secretions in pediatric subjects

SUMMARY:
Children's tear film and ocular surface are increasingly exposed to environmental factors. The tear film is the most important barrier protecting the eye from external insults such as pollen, dust, sand. If a foreign substance is not washed away by the tear film, it eventually reaches the ocular surface resulting in eye irritation, ocular secretions, and/or allergic response. Primary intervention is aimed at avoiding allergens and using eye lubricants to facilitate the washout of the foreign substance. It is also recommended to regularly clean the children's eyes to avoid infections. Topical medications are usually recommended only in the presence of infectious conjunctivitis.

Ocular secretions are also commonly observed in newborn babies. Neonatal ocular discharge is often related to congenital nasolacrimal duct obstruction (CNLDO) which normally occurs within the first weeks of age. CNLDO (also known as dacryostenosis) results from a congenital abnormality of the lacrimal drainage system in the form of a membranous obstruction of the nasolacrimal duct of one or both eyes. In most cases, blocked tear ducts open spontaneously within the first 6-12 months of age. Traditionally, management of CNLDO consists of frequent lacrimal sac massages and regular cleaning of the eyes. Topical antibiotic therapy is indicated only with the clinical evidence of infection.

For these reasons, an interventional, non-comparative, single-center Post Marketing Clinical Follow-up (PMCF) study was planned to evaluate the performance and safety of "LUXIDROPIN BABY & JUNIOR" used to facilitate the removal of ocular secretions in pediatric subjects.

The objectives of the PMCF study are confirmation of the performance, collection of additional safety data regarding expected adverse events and detection of potential unexpected adverse events associated with the use of "LUXIDROPIN BABY & JUNIOR" according to the Instructions for Use (IFU).

Each pediatric subject whose parent(s)/legal guardian signed an Informed Consent Form (ICF), will enter the screening and baseline phase (the 2 visits will coincide) during which baseline procedures will be completed.

At baseline visit (V0), "LUXIDROPIN BABY & JUNIOR" will be administered to the enrolled subject.

The patient will perform 2 on-site visits: V0 and V2/EOS. To monitor the safety, 1 phone contact is planned (V1) to check for potential adverse events and concomitant medications intake.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric subjects whose ICF will be signed by parent(s) or legal guardian;
* M & F newborns (10-27 days), infants (28 days-23 months), children (2-11 years);
* Ocular discharge (pediatric subjects presenting with ocular secretions due nasolacrimal duct obstruction; pediatric subjects presenting with amblyopia, redness of the ocular mucosa, burning, itching due to climatic factors or seasonal allergies).
* Willingness not to use other ophthalmic solutions (spray or drops) during the entire study.

Exclusion Criteria:

* Preterm newborns;
* Pediatric subjects with congenital abnormalities of the eye, physical trauma, corneal infiltrate or ulcers in either eye. Presence of any relevant organic, systemic or metabolic disease (particularly significant history of cardiac, renal, neurological, psychiatric, oncology, endocrinology, metabolic or hepatic disease), or abnormal laboratory values that will be deemed clinically significant based on predefined values;
* Pediatric subjects with/without eye infections requiring treatment with topical or systemic antibiotics;
* Previous eye surgery;
* Suspected other - different - eyes clinical conditions (e.g. glaucoma);
* Suspected known hypersensitivity or allergy to Investigational Product (IP) components;
* Other clinically significant and uncontrolled pathologies that may interfere with study results (e.g. diabetes);
* Participation in another investigational study;
* Parent(s)' and/or patients' inability to follow all study procedures, including attending all site visits, tests and evaluations;
* Parent(s)' and/or patients' mental incapacity that precludes adequate understanding or cooperation.

Ages: 10 Days to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with clinical resolution, measured as the absence of ocular secretions, will be assessed at the end of the study visit (Day 4). | From baseline (Day 0) to 4 days (Day 4 (96h))

SECONDARY OUTCOMES:
To evaluate the performance of "LUXIDROPIN BABY & JUNIOR" to relieve redness of the ocular mucosa and itching, through Visual Analogue Scale (VAS( for assessment of ocular discomfort | From baseline (Day 0) to 4 days (Day 4 (96h))
  Visual Analogue Scale:
  Minimum value = 0; Maximum value = 10; Higher scores mean a better outcome.
To evaluate the safety and tolerability of "LUXIDROPIN BABY & JUNIOR" through eye examination and assessment of AEs including the relationship of the AE to the IP (e.g. local allergic reaction) | From baseline (Day 0) to 2 days (Day 2 (48 h)) and 4 days (Day 4 (96h))
To evaluate the capability of "LUXIDROPIN BABY & JUNIOR" to improve the quality of life (QoL), through Visual Analogue Scale (VAS) for assessment of the QoL | End of study visit (Day 4 (96h))
  Visual Analogue Scale:
  Minimum value = 0; Maximum value = 10; Higher scores mean a better outcome
To evaluate the parent(s) or children's satisfaction through a Rensis Likert 5 points patients satisfaction scale | End of study visit (Day 4 (96h))
  Rensis Likert 5 points patients satisfaction scale Minimum value: Very dissatisfied Maximum value: Very satisfied Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Policlinico Mater Domini - Università Magna Grecia di Catanzaro, Catanzaro, CZ, Italy